CLINICAL TRIAL: NCT06941857
Title: A Phase 2 Study of NC410 and FOLFIRINOX in Combination With Nivolumab With or Without Ipilimumab in Patients With Treatment-naïve, Metastatic Pancreatic Cancer
Brief Title: NC410 and FOLFIRINOX in Combination With Nivolumab With or Without Ipilimumab in Patients With Untreated Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: NextCure, Inc. (Industry); Lustgarten Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J2541; IRB00486324 (Other: Johns Hopkins Medical Institution)
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer
Keywords: Nivolumab; Ipilimumab; NC410 (NextCure LAIR-2 (Leukocyte-Associated Immunoglobulin-like Receptor-2) fusion protein); Oxaliplatin; Irinotecan; Folinic Acid; 5-Fluorouracil; Folfirinox; Immunotherapy; Anti-PD-1 (anti-check point inhibitor); PD-L1 (check point inhibitor); Anti-CTLA-4 (anti-cytotoxic T-lymphocyte-associated antigen 4); Metastatic Pancreatic Cancer; Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma (PDAC); Carcinoma; Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma | interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 - FOLFIRINOX/NC410/Nivolumab (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: Folinic Acid; Drug: 5-Fluorouracil (5-FU); Drug: NC410; Drug: Nivolumab
- Arm 2 - FOLFIRINOX/NC410/Nivolumab/Ipilimumab (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: Folinic Acid; Drug: 5-Fluorouracil (5-FU); Drug: NC410; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Oxaliplatin — 65mg/m2 will be administered as a 120 minute IV Infusion (-10/+ 20 minutes) on day 1 of each cycle every 2 weeks. Each cycle length is 14 days. The two arms will enroll sequentially (starting with Arm 1 followed by Arm 2).
Drug: Irinotecan — 150 mg/m2 will be administered as a 90 minute IV Infusion (-10/+ 20 minutes) on day 1 of each cycle every 2 weeks. Each cycle length is 14 days. The two arms will enroll sequentially (starting with Arm 1 followed by Arm 2).
Drug: Folinic Acid — 50 mg will be administered as a 15 minute IV infusion (-5/+20 min) on day 1 of each cycle every 2 weeks. Each cycle length is 14 days. Folinic acid can be given concurrent with irinotecan. The two arms will enroll sequentially (starting with Arm 1 followed by Arm 2).
Drug: 5-Fluorouracil (5-FU) — 2400 mgm2 will be administered as a continuous IV Infusion (-120/+ 120 minutes) over approximately 46 hours on day 1 of each cycle every 2 weeks. Each cycle length is 14 days. The two arms will enroll sequentially (starting with Arm 1 followed by Arm 2).
Drug: NC410 — 100 mg will be administered as a 60 minute IV Infusion (-10/+ 20 minutes) on day 1 of each cycle every 2 weeks. Each cycle length is 14 days. The two arms will enroll sequentially (starting with Arm 1 followed by Arm 2).
  Other Names: NextCure LAIR-2 fusion protein
Drug: Nivolumab — 400 mg will be administered as a 30 minute IV Infusion (-5/+20 minutes) once on Cycle 1 Day 1. Each cycle length is 14 days. The two arms will enroll sequentially (starting with Arm 1 followed by Arm 2).
  Other Names: OPDIVO
Drug: Ipilimumab — 50 mg will be administered as a 30 minute IV Infusion (-5/+20 minutes) once on Cycle 1 Day 1. Each cycle length is 14 days. The two arms will enroll sequentially (starting with Arm 1 followed by Arm 2).
  Other Names: YERVOY
  Arms: Arm 2 - FOLFIRINOX/NC410/Nivolumab/Ipilimumab

SUMMARY:
The purpose of this study is to evaluate safety of the treatment regimen and identify any novel toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1.
* Metastatic histologically or cytologically confirmed pancreatic ductal adenocarcinoma.
* Have metastatic disease
* Must not have received prior systemic treatment for pancreatic cancer.
* Have measurable disease based on RECIST 1.1.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests and procedures.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test.
* For both Women and Men, must use acceptable form of birth control while on study.
* Must understand the study regimen, its requirements, risks and discomforts and is able and willing to sign the informed consent form in accordance with regulatory and institutional guidelines.

Exclusion Criteria:

* Have had prior chemotherapy for pancreatic cancer or prior chemotherapy within 5 years of enrollment for other cancer diagnoses.
* Has received radiotherapy for pancreatic cancer.
* Are receiving or have received any investigational agent or used an investigational device within 28 days prior to Day 1 of treatment in this study.
* Has undergone major surgery, other than diagnostic surgery (i.e. surgery done to obtain a biopsy for diagnosis or an aborted Whipple), within 28 days prior to Day 1 of treatment in this study.
* Is expected to require any other form of systemic or localized antineoplastic therapy while on study.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4, or anti-Lag-3 antibodies.
* Has received a live vaccine or live-attenuated vaccine within 28 days prior to the first dose of study drug.
* Prior tissue or organ allograft regardless of need for immunosuppression, including corneal allograft.
* Has uncontrolled acute or chronic medical illness.
* Has history of central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has known additional malignancy that is progressing and requires active treatment.
* Has active autoimmune disease.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Requirement for daily supplemental oxygen.
* History of interstitial lung disease, non-infectious pneumonitis or uncontrolled lung diseases including pulmonary fibrosis, acute lung diseases, chronic obstructive pulmonary disease (COPD), asthma requiring medication, etc.
* Known history of human immunodeficiency virus (HIV).
* Active or chronic hepatitis B or hepatitis C.
* Unable to undergo venipuncture and/or tolerate venous access.
* Has known psychiatric or substance use disorder that would interfere with cooperation with the requirements of the trial.
* Pregnant or breastfeeding
* A WOCBP who has a positive urine pregnancy test within 72 hours prior to study drug initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing unexpected toxicities. Unexpected toxicities are toxicities related to the study drug required treatment discontinuation. | 4 years
  When calculating the incidence of Adverse Events (AEs), each AE (as defined by NCI CTCAE v5.0) will be counted only once for a given subject.

SECONDARY OUTCOMES:
Progression- Free Survival (PFS) | 4 years
  PFS is defined as the number of months from the date of first dose to disease progression (PD as assessed using RECIST 1.1 criteria) or death due to any cause. PFS will be censored at the date of the last scan for subjects without documentation of disease progression at the time of analysis. PFS will be censored at time of first dose for patients that do not have a follow-up scan. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30percent decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20percent increase in sum of diameters of target lesions, Stable Disease (SD) is <30percent decrease or <20percent increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Response Rate (ORR) | 4 years
  ORR is defined as the number of subjects with PR or CR according to RECIST 1.1. Subjects who discontinue due to toxicity or clinical progression prior to post-baseline tumor assessments will be considered as non-responders. CR = disappearance of all target lesions, PR is =>30percent decrease in sum of diameters of target lesions, progressive disease (PD) is >20percent increase in sum of diameters of target lesions, stable disease (SD) is <30percent decrease or <20percent increase in sum of diameters of target lesions.
Disease Control Rate (DCR) | 4 years
  DCR is defined as the number of subjects achieving stable disease or better (SD, PR or CR) according to RECIST 1.1. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30percent decrease in sum of diameters of target lesion, Stable Disease (SD) is <30percent decrease or <20percent increase in sum of diameters of target lesions.
Overall Survival (OS) | 4 years
  OS is defined as the number of months from the date of first dose until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bever, MD, Principal Investigator — SKCCC Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No